CLINICAL TRIAL: NCT04630496
Title: Pre-Operative Exercise Challenge In Geriatric Thoracic Patients
Brief Title: Geriatric Thoracic Surgery Ambulation Challenge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Michael Jaklitsch, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-061
Record Dates: First submitted 2020-11-13; First posted 2020-11-16 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Thoracic Diseases; Surgery; Therapy, Exercise
Keywords: Thoracic Diseases; Lung Resection; Perioperative activity; Pedometer tracker
MeSH Terms: conditions — Thoracic Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRE-OPERATIVE EXERCISE TRACKING (Experimental): Participant baseline information will be collected from their electronic medical records.
  After enrollment, participants will be provided a mobile device (Fitbit) to wear for tracking steps for 1 week prior to their scheduled surgery.
  Participants will keep a log of daily steps for the 1 week they are wearing the device and receive one progress check-in call during the week.
  The device and log will be turned in either on a pre-surgery clinic visit or on the day of surgery whichever comes first.
  Interventions: Behavioral: Fitbit

INTERVENTIONS:
Behavioral: Fitbit — Electronic activity tracker
  Other Names: mobility tracker; pedometer

SUMMARY:
This study is examining collecting data on steps walked (ambulation) per day by thoracic surgery patients over the age of 65 years-old before surgery.

The name(s) of the study device involved in this study is:

* Fitbit inspire

DETAILED DESCRIPTION:
This research study is a Feasibility Study, which is the first-time investigators are examining the use of a Fitbit by thoracic surgery patients over the age of 65 years-old before surgery. The study is looking to see if patients can wear a wrist step-tracker and keep a log of their daily step counts for one week. The study is looking to see if people are willing to keep track of their daily steps, so in the future participants may be provided with step-goals to achieve and their steps prior to surgery can be accurately measured.

This research study involves using a Fitbit tracker to record daily steps over the course of 1 week prior to scheduled surgery. Participants will be given a step tracker in clinic and instructed on its use. During the 1 week period, participants will be called by a study team to check on progress.

After a week, participants will be asked to return the step-tracker and their log either at a scheduled pre-surgery clinic visit or in the pre-operative area which ever comes first.

It is expected that about 30 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Patients Aged ≥ 65 years

  * Who are preparing to undergo thoracic surgery at Brigham and Women's Hospital (BWH)

Exclusion Criteria:

* Patients who are completely non-ambulatory (i.e. wheelchair-bound-patients) *
* Those who lack capacity to consent due to cognitive disease.
* Patient for which surgery is felt to be more urgent and therefore performed earlier then our required timeframe for intervention.
* Patients with cardiac disease or angina for which formal cardiac testing is required for clearance.

  * Our exclusion criteria do not include patients with gait disturbances or those who require assistance devices for ambulation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Step Tracking Rate | 1 week
  Feasibility will be determined by the successful tracking of steps and keeping a diary of step-count for one-week duration. Completion of a minimum of 5/7 days will be considered as a success
Diary of Steps Rate | 1 week
  Feasibility will be determined by the successful tracking of steps and keeping a diary of step-count for one-week duration. We will consider completion of a minimum of 5/7 days as a success.
Return Rate | 1 week
  If 90% of trackers are returned, it will be considered a successful return.
Data Retrieval Rate | 1 week
  assess extraction of the data from the mobility upon return. Success will be considered if 90% of data is retrievable

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Jaklitsch, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation